CLINICAL TRIAL: NCT04681560
Title: The Effect of Polychemotherapy on Endothelial Function Ans Vessel Age in Cancer Patients.
Brief Title: Impact of Platinum-based Cancer Treatment on Endothelial Function
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 1019
Record Dates: First submitted 2020-04-18; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2019-09

CONDITIONS: High Blood Pressure; Cardiovascular Complication
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this research we investigate endothelial function in cancer patients who received platinum based chemotherapy.

DETAILED DESCRIPTION:
The goal of the study is to evaluate endothelial function in patients with platinum-based versus non-platinum-based chemotherapy.

Endothelial function was evaluated via Angioscan( the apparatus that evaluate the stiffness of vessels by pulse wave velocity) and serum levels of endothelial nitric oxide synthase (ENOS),endothelin1.

Patients with gastrointestinal, ovarian, bladder and brest cancer would be included.

Patients with malignancies were followed-up from 2 weeks to 3 month after start of chemotherapy, Medical records and hospital databases were searched for all the patients treated with different chemotherapy treatment for any kind of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subject has solid cancer
* Subject is expected to start chemotherapy

Exclusion Criteria:

* Pregnancy and lactation
* Severe impaired kidney function
* Severe hepatic impairment
* Mental disease
* Acute myocardial infarction 28 days ago or earlier
* Acute Cerebrovascular Event 1 month ago or earlier
* Rhythm disturbance that complicate pulse wave velocity evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study included 60 patients, that have diagnosis solid cancer of any stage and localisation.All of them is expected to start platinum based or non platinum based chemotherapy.The study proseeds in Chemotherapy department at City Hospital No.1.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of blood pressure | Before start of chemotherapy (1 hour after including in the trial)
  Both systolic and diastiolic blood pressure were measured in the office in the seated position, noninvasively.
Evaluation of flow-mediated vasodilation and pulse-wave velocity | Before start of chemotherapy (1 hour after including in the trial)
  Flow-mediated dilatation and pulse-wave velocity were measured via "Angioscan" apparatus in the seated position.The cuff inflation period of 5 min was initially decided to produce adequate hyperaemia to allow flow-mediated dilatation. The scanning period used in our trial was 1 minite before and 9 minutes after the cuff deflation.
Evaluation of concetration of ENOS and Big Endothelin in blood sampling | Before start of chemotherapy (1 hour after including in the trial)
  Blood was collected from the cubital vein to 10.0 ml/ 6.0 ml red top tubes (without clot activator). The sample was then separated by centrifugation. The serum was frozen to -20C.

SECONDARY OUTCOMES:
Evaluation of blood pressure | In range of 3 -12 weeks after start of chemotherapy (before next chepotherapy drug injection)
  Both systolic and diastiolic blood pressure was measured in the office in the seated position, noninvasively.
Evaluation of flow-mediated vasodilation and pulse-wave velocity | In range of 3 -12 weeks after start of chemotherapy (before next chepotherapy drug injection)
  Flow-mediated dilatation and pulse-wave velocity were measured via "Angioscan" apparatus in the seated position.The cuff inflation period of 5 min was initially decided to produce adequate hyperaemia to allow flow-mediated dilatation. The scanning period used in our trial was 1 minite before and 9 minutes after the cuff deflation.
Evaluation of concetration of ENOS and Big Endothelin of blood sampling | In range of 3 -12 weeks after start of chemotherapy (before next chepotherapy drug injection)
  Blood was collected from the cubital vein to 10.0 ml/ 6.0 ml red top tubes (without clot activator). The sample was then separated by centrifugation. The serum was frozen to -20C.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Shchekochikhin, PhD, Principal Investigator — I.M. Sechenov First Moscow State Medical University
Locations (2):
- Russia (2):
  - Olga Andreeva, Moscow
  - First Moscow State Medical University., Moscow